CLINICAL TRIAL: NCT02313519
Title: A Randomized Clinical Study of the Efficacy of a Formulation of Four Probiotics for the Prevention of Post-operative Complications in Patients Undergoing Colorectal Surgery
Brief Title: Probiotics in the Prevention of Complications After Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Evangelos J. Giamarellos-Bourboulis, M.D. (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor-Investigator, Evangelos J. Giamarellos-Bourboulis, M.D., Associate Professor of Medicine, University of Athens
Organization: University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LACT002
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Postoperative Complications
Keywords: Infections; anastomotic leakage
MeSH Terms: conditions — Postoperative Complications; Infections; Anastomotic Leak | interventions — Probiotics; Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Capsules of powdered glucose polymer given one capsule every 12 hours for 15 days
  Interventions: Dietary Supplement: Placebo
- Probiotics (Active Comparator): Capsules containing Lactobacillus acidophilus LA-5 [1.75x10^9 cfu], Lactobacillus plantarum [0.5x10^9 cfu], Bifidobacterium lactis BB-12 [1.75x10^9cfu], and Saccharomyces boulardii [1.5x10^9] per capsule. One capsule is given every 12 hours for 15 days
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Probiotics are prepared in capsule form
  Other Names: Lactobacillus, Bifidobacterium and Saccharomyces boulardii
  Arms: Probiotics
Dietary Supplement: Placebo — Glucose powder
  Other Names: Placebo capsules
  Arms: Placebo

SUMMARY:
Based on the need of large-scale, trials to explore the use of probiotics to reduce post-operative complication rate, a randomized controlled trial is designed to investigate the impact of a probiotics treatment protocol on postoperative morbidity in an open elective colonic surgery cohort. The major objective is reduction of post-operative complications after 30 days.

DETAILED DESCRIPTION:
Major colorectal surgery, i.e. surgery involving a wide colon resection and/or a very low anastomosis, remains problematic, despite great advances in medico-pharmaceutical treatment, improvement in surgical techniques, and sophisticated postoperative management. Such surgery is still accompanied by an unacceptably high morbidity of 15% to 23.2% leading to an increase in the number of ventilatory support days, prolongation of total hospital stay, significantly higher medical costs, patient suffering, and, unfortunately mortality. Worse than this, nowadays, infections and sepsis are by far the most common morbidities, either as initial cause or as a consequence of another complication, such as anastomotic leakage. Ongoing clinical studies have reported probiotic therapies to be beneficial in elective surgery cases, since they have been shown to successfully modulate the GI flora in a plethora of medical settings and in critically ill and trauma patients. More precisely, recent randomized controlled studies and meta-analyses in elective surgery and abdominal surgery patients have demonstrated that the perioperative use of probiotics is safe and reduces both the incidence of postoperative wound infections, sepsis, post-operative pneumonia and other infections, and the necessary duration of hospital stay and length of antibiotic therapy. However, there exist few controlled, large-scale, trials comparing the current standard treatment with the probiotic concept and showing the superiority of the latter in colonic surgery with regard to a reduced complication rate. Therefore, the investigators decided to conduct a randomized controlled trial to investigate the impact of a probiotics treatment protocol on postoperative morbidity in an open elective colonic surgery cohort. The major objective is to evidence a reduction in 30-day infectious, surgery-related morbidity: any surgical site infection; organ specific infections; systemic infections and anastomotic leakage. Minor objectives related to the reduction in other non-infectious complications, as well as the assessment of outcome indicators such as the number of days in postoperative ileus, on mechanical ventilation, stay in ICU, total hospitalization and mortality in the 30-day post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Acceptable nutritional status and programmed for open surgery for colorectal cancer.
* Operation by the same consultant either as surgeon or as the primary assistant.

Exclusion Criteria:

* Inability to provide written informed consent
* The need only for emergency or palliative surgery
* American Society of Anaesthesiologists (ASA) class of IV
* Pregnancy or lactation
* Inflammatory bowel disease
* Use of antibiotics during the last 10 days before surgery
* Recent steroid therapy or preoperative neoadjuvant chemotherapy or radiotherapy
* Pre-existing signs of bacterial [white cell count, body temperature] or viral infection [hepatitis B or C, human immunodeficiency virus, cytomegalovirus].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  The total of postoperative complications observes in each study group. These comprise: any anastomotic leakage; abdominal wound infection and dehiscence; organ specific infections, such as pneumonia, urinary tract and central vein port-site infections, and systemic infections [bacteraemia, fungal infections] as regularly defined by positive cultures, radiograms, increased white blood cell count or purulent material discharge; sepsis and septic shock

SECONDARY OUTCOMES:
Minor complications | 30 days
  Rate of minor events in each group. These comprise peripheral vein thrombosis or pulmonary embolism and cardio-pulmonary or renal insufficiency. Moreover, the number of days on mechanical ventilation, in postoperative ileus, of total hospitalization, as well as 30-day mortality is taken into account.
Cytokine levels | 4 days
  Measurement of serum cytokines in subgroups of patients
Cytokine gene transcripts | 4 days
  Measurement of gene transcripts in whole blood in subgroups of patients

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Kotxampassi, MD, PhD, Study Chair — AXEPA University of Thessaloniki, 1st Department of Propedeutic Surgery, Thessaloniki, Greece; Evangelos Giamarellos-Bourboulis, MD, PhD, Principal Investigator — University of Athens, 4th Department of Internal Medicine, Athens, Greece

REFERENCES:
- [Background] Giamarellos-Bourboulis EJ, Bengmark S, Kanellakopoulou K, Kotzampassi K. Pro- and synbiotics to control inflammation and infection in patients with multiple injuries. J Trauma. 2009 Oct;67(4):815-21. doi: 10.1097/TA.0b013e31819d979e. PMID 19820590
- [Background] Kotzampassi K, Giamarellos-Bourboulis EJ, Voudouris A, Kazamias P, Eleftheriadis E. Benefits of a synbiotic formula (Synbiotic 2000Forte) in critically Ill trauma patients: early results of a randomized controlled trial. World J Surg. 2006 Oct;30(10):1848-55. doi: 10.1007/s00268-005-0653-1. PMID 16983476
- [Derived] Kotzampassi K, Stavrou G, Damoraki G, Georgitsi M, Basdanis G, Tsaousi G, Giamarellos-Bourboulis EJ. A Four-Probiotics Regimen Reduces Postoperative Complications After Colorectal Surgery: A Randomized, Double-Blind, Placebo-Controlled Study. World J Surg. 2015 Nov;39(11):2776-83. doi: 10.1007/s00268-015-3071-z. PMID 25894405